CLINICAL TRIAL: NCT03626935
Title: 3D Printed Customized Guide in Ankle Arthrodesis
Brief Title: 3D Printed Guide in Ankle Arthrodesis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Xiaojun Duan, Deputy Director of the Center for Joint Surgery, Southwest Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 3DAnkleGuide
Record Dates: First submitted 2018-08-08; First posted 2018-08-13 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Ankle Injuries
Keywords: ankle joint; arthrodesis; 3d printing; customized guide
MeSH Terms: conditions — Ankle Injuries; Ankylosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3D-printed customized guide plate (Experimental): 3D-printed customized guide plate will be used to guide the Kirschner wires in ankle arthrodesis.
  Interventions: Device: 3D-printed customized guide plate

INTERVENTIONS:
Device: 3D-printed customized guide plate — 3D-printed customized guide plate will be used in the ankle arthrodesis to help reduce operation time and reduce intra-operative radiation.

SUMMARY:
This study applies 3D-printed customized guide plate in assisting the accurate drilling of Kirschner wire in ankle arthrodesis. This technique can shorten the operation time, reduce the intra-operative radiation, and do not affect the surgical outcome.

DETAILED DESCRIPTION:
Ankle arthrodesis is the standard procedure for treating end-stage joint diseases. In order to improve the surgical outcome and reduce the operation time, 3D-printed customized guide plates are fabricated using patients' ankle DICM data of ankle via CT examinations. Two 2mm Kirschner wires are drilled with the help of the guides; the C-arm fluoroscopy is used to confirm the position of the wires before applying the cannulated screws for effective fixation.

In the past when there were no customized guides, the surgeons would drill the Kirschner wire according to his/her previous experience and then use C-arm fluoroscopy to confirm whether the position of the wire is satisfactory; if not, repeated procedure will be performed. This would lead to an increase in the duration of surgery and intra-operative radiation, which is detrimental to both the surgeon and the patient. This problem is well solved by applying the 3D-printed customized guides.

The application procedure for the customized guide plates: the model of the ankle joint is established according to the patient's CT scan data to prepare the customized guide plate, then sterilize them for future use. Apply routine surgical treatment to the ankle joint surface, reset the fusion joint to the functional position, and drill two 2mm Kirschner wires with the guidance of the guide plate. If the locations of the fusion joint and the Kirschner wires are satisfactory under the C-arm fluoroscopy, drill the cannulated screws for final fixation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who receive ankle arthrodesis and consider internal fixation with screws

Exclusion Criteria:

* Patients who receive ankle arthrodesis but do not consider internal fixation with screws

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
Operation time | Intraoperative
  Operation time for internal fixation

SECONDARY OUTCOMES:
Postoperative ankle AOFAS scale | Postoperative 1,6,12 months
  Postoperative American Orthopaedic Foot and Ankle Society (AOFAS) Scale of the ankle joint. Scale range: 0-100 points. Outcome evaluation: Excellent, 90-100; Good, 75-89; Average, 50-74；Poor, <50.
Fusion rate | Postoperative 1,6,12 months
  Fusion rate of the ankle joint

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Duan, M.D., Principal Investigator — Southwest Hospital, China
Locations (1):
- Southwest Hospital, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Derived] Duan X, He P, Fan H, Zhang C, Wang F, Yang L. Application of 3D-Printed Personalized Guide in Arthroscopic Ankle Arthrodesis. Biomed Res Int. 2018 Sep 12;2018:3531293. doi: 10.1155/2018/3531293. eCollection 2018. PMID 30276205